CLINICAL TRIAL: NCT01196585
Title: ULTRASONOGRAPHY GUIDED PLEURAL NEEDLE BIOPSY VERSUS COMPUTED TOMOGRAPHY GUIDED ABRAMS PLEURAL NEEDLE BIOPSY FOR DIAGNOSIS OF PATIENTS WITH PLEURAL EFFUSIONS: A RANDOMIZED CONTROLLED TRIAL
Brief Title: Ultrasonography Guided Pleural Biopsy Versus Computed Tomography Guided Pleural Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Muzaffer Metintas, ESOGU Medical Faculty Department of Chest Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 082010/2
Record Dates: First submitted 2010-08-26; First posted 2010-09-08 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-09

CONDITIONS: Pleural Diseases
Keywords: Pleura; biopsy; diagnosis; CT; ultrasonography
MeSH Terms: conditions — Pleural Diseases; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients under CT- guided pleural biopsy (Experimental): Arm A: Patients who go under CT-guided pleural needle biopsy for pleural diseases
  Interventions: Procedure: CT-Guided pleural needle biopsy with Abrams' needle
- Patients under ultrasonography guided needle biopsy (Experimental): Arm B: Patients who go under ultrasonography guided cutting needle pleural biopsy for pleural diseases
  Interventions: Procedure: Ultrasonography guided cutting pleural needle biopsy

INTERVENTIONS:
Procedure: CT-Guided pleural needle biopsy with Abrams' needle — Patients will be randomized into two groups: Group A: CT-guided Abrams' needle biopsy.
  Arms: Patients under CT- guided pleural biopsy
Procedure: Ultrasonography guided cutting pleural needle biopsy — Patients will be randomized into two groups: Group B: Ultrasonography guided cutting-needle biopsy.
  Arms: Patients under ultrasonography guided needle biopsy

SUMMARY:
This study aims to compare the diagnostic efficiency and reliability of Abrams' needle pleural biopsy under computerized tomography guidance with that of cutting-needle pleural biopsy under ultrasonography guidance in patients with pleural effusion.

DETAILED DESCRIPTION:
Background. In cases with pleural effusion, tissue samples can be obtained through Abrams' needle pleural biopsy, thoracoscopy, or cutting-needle pleural biopsy under the guidance of computerized tomography or ultrasonography for histopathological analysis. This study aims to compare the diagnostic efficiency and reliability of Abrams' needle pleural biopsy under computerized tomography guidance with that of cutting-needle pleural biopsy under ultrasonography guidance in patients with pleural effusion.

Methods. Patients with exudative pleural effusion, who could not be diagnosed by cytological analysis, will be included in the study. All patients were randomized following the thoracic computerized tomography with contrast enhancement. Patients either underwent Abrams' needle pleural biopsy under computerized tomography guidance or the cutting-needle pleural biopsy under ultrasonography. The two groups will be compared in terms of diagnostic efficiency and in terms of complications associated with the methods used.

ELIGIBILITY:
Inclusion Criteria:

* Patients with exudative pleural effusion who require invasive procedure for diagnosis

Exclusion Criteria:

* Patients without pleural effusion

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To compare the sensitivities and specificities of two diagnostic methods for pleural diseases to establish which method is more effective. | 28-months
  The investigators will determine which method more efficient for the diagnosis of pleural diseases establishing sensitivity and specificity of the methods. After establishment of sensitivity, specificity and side effects for each diagnostic method the investigators will compare them according to the method and determine which method is more efficient.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability. | 28-months
  All patients in both arm will be followed for complications of the diagnostic method. Complications experienced by the patients will be determined and recorded in special forms. Each complication will be measured with own characteristic such as pain, local infection, pneumothorax,local inavsion of disease, haemoragy etc.

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffer Metintas, Professor, Principal Investigator — ESOGU Medical Faculty
Locations (1):
- Eskisehir Osmangazi University Medical Faculty department of Chest Diseases, Eskişehir, Turkey (Türkiye)

REFERENCES:
- [Background] Metintas M, Ak G, Dundar E, Yildirim H, Ozkan R, Kurt E, Erginel S, Alatas F, Metintas S. Medical thoracoscopy vs CT scan-guided Abrams pleural needle biopsy for diagnosis of patients with pleural effusions: a randomized, controlled trial. Chest. 2010 Jun;137(6):1362-8. doi: 10.1378/chest.09-0884. Epub 2010 Feb 12. PMID 20154079